CLINICAL TRIAL: NCT04110769
Title: Development of Biomarker for the Evaluation of Response After Neoadjuvant Therapy in Patients With Pancreatic Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Song Cheol Kim, Professor, Asan Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: NACTMarker-01
Record Dates: First submitted 2019-08-23; First posted 2019-10-01 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Genetic Change; Chemotherapy Effect; Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Responders (Experimental): The investigator will administer neoadjuvant chemotherapy After neoadjuvant chemotherapy, multidisciplinary team will decide to surgery or continuing chemotherapy based on following imaging studies and tumor markers.
  The patients who undergo surgery after neoadjuvant chemotherapy will be included responders.
  Interventions: Diagnostic Test: next generation sequencing
- Non-responders (Active Comparator): The patients who show cancer progression even after neoadjuvant chemotherapy will be classify with non-responder. And the investigator will change palliative chemotherapy.
  Interventions: Diagnostic Test: next generation sequencing; Diagnostic Test: following next generation sequencing

INTERVENTIONS:
Diagnostic Test: next generation sequencing — the investigator will compare genetic mutation between responder and non-responder using next generation sequencing examination.
Diagnostic Test: following next generation sequencing — The patient will be examined next generation sequencing before changing palliative chemotherapy for non-responders.
  Arms: Non-responders

SUMMARY:
The purpose of this study is to identify and apply biomarkers that can provide better information than previous imaging and blood tests when evaluating the response after neoadjuvant chemotherapy in pancreatic cancer patients who require neoadjuvant therapy before surgery.

DETAILED DESCRIPTION:
BACKGROUND

* Pancreatic cancer is a rare cancer of the digestive system, but it is known to have a poor prognosis with a very poor survival rate. Five-year survival rate of all patients with pancreatic cancer is less than 6%, and only 10-20% of patients are eligible for surgery at the time of diagnosis.
* Postoperative complications of pancreatic cancer are reported in 30-50% of cases, and only 50% of patients undergoing postoperative chemotherapy at the appropriate time after surgery are reported. As a result of these concerns, the study of neoadjuvant chemotherapy (NACT) was begun. Recently, several clinical studies of chemotherapy have been performed. Cancer (BRPC), locally advanced pancreatic cancer (LAPC) patients who have had difficult surgical resection, are turning to treatment by combining surgical treatment after NACT.
* Although standard treatments for advanced chemotherapy have yet to be established through many clinical studies, the most commonly used regimens are FOLFIRINOX (fluorouracil, leucovorin, irinotecan, and oxaliplatin), gemcitabine and nab-paclitaxel. The response rate after prior chemotherapy is known as 30-50%, and the response of patients undergoing surgery after prior chemotherapy was compared with the serum markers before and after chemotherapy through CA19-9, PET-CT, and CT. The response could be estimated by the reduction, the size change in the imaging test, or the decrease in SUVmax. However, there are only a few studies on genetic and molecular studies of which patients will respond. Under these circumstances, this study on the discovery of biomarkers for the response of advanced chemotherapy in patients with pancreatic cancer may provide guidelines for the application of advanced chemotherapy and the selection of appropriate drugs, as well as clues for future research.

Primary endpoint:

-Discovery of genetic mutation in response to NACT

METHODOLOGY Recruitment and sample collection of patients undergoing NACT Identifying pancreatic cancer specific candidate genes in response to NACT

EXPECTED RESEARCH RESULTS

* Predictable genes and biomarkers of responsiveness for NACT can be identified.
* It is possible to understand the progress of pancreatic cancer widely
* The development of biomarkers that can predict the response of NACT
* In patients with BRPC or LAPC who need NACT, appropriate screening will be possible.

ELIGIBILITY:
Inclusion Criteria:

* The patients who are going to administer neoadjuvant chemotherapy for borderline resectable or locally advanced pancreatic cancer
* Performance: 0-2
* No distant metastasis
* Patients who consented to and signed the consent

Exclusion Criteria:

* Distant metastasis
* Patients included in other clinical studies that may affect this study
* Patients who cannot follow the directions of the researcher
* Patients with moderate or severe comorbidities who are thought to have an impact on quality of life or nutritional status (cirrhosis, chronic kidney failure, heart failure, etc.)
* Pelvic tumor, benign tumor, malignant tumor in other organs
* Patients who received prior chemotherapy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-07-17 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
The rate of genetic mutation | before neoadjuvant chemotherapy
  Discovery of genetic mutation in response to neoadjuvant chemotherapy

SECONDARY OUTCOMES:
oncologic outcome | 3 - 5 years after surgery
  overall survival and recurrence free survival

CONTACTS AND LOCATIONS:
Overall Officials: Song-Choel Kim, MD.PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan medical center, Seoul, South Korea